CLINICAL TRIAL: NCT04326595
Title: Histopathological Evaluation of Product of Conception in Sporadic and Recurrent Abortions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MOHAMMED HAGGAG HASHIM, Principal Investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: histopathology in abortion
Record Dates: First submitted 2020-03-25; First posted 2020-03-30 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Recurrent Abortion
MeSH Terms: conditions — Abortion, Habitual | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: 1. Full detailed history taking .
  2. Through clinical examination .
  3. pregnancy was confirmed by ultrasound examination or serum beta human chorionic gonadotropins (β-HCG) level for patients.
  4. All patients had routine laboratory tests including blood group, Rh factor, complete blood count, and electrolytes.
  5. Then the all tissues obtained at evacuation should be submitted for histopathological examination
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical termination (Active Comparator)
  Interventions: Procedure: surgical and medical evacuation
- medical termination (Active Comparator)
  Interventions: Procedure: surgical and medical evacuation

INTERVENTIONS:
Procedure: surgical and medical evacuation — surgical evacuation:the dilation of the cervix and surgical evacuation of the uterus (potentially including the fetus, placenta and other tissue) medical evacuation: induction of abortion by the use of ecbolics

SUMMARY:
1. To evaluate histopathological findings of products of conception in both sporadic and recurrent miscarriage.
2. To determine the prevalence of chronic histiocytic intervillositis in both sporadic and recurrent miscarriage.

DETAILED DESCRIPTION:
Early miscarriage is a term used to describe the loss of pregnancy within the first 12 weeks of gestation .This diagnosis concerns 10-15% of all pregnancies and is made based on additional tests such as serial determinations of chorionic gonadotropin concentration and imaging examinations ultrasonography. Depending on the clinical presentation and results of ultrasonography, miscarriages can be divided into complete spontaneous miscarriage, and incomplete miscarriage, when the width of the echo of residual tissues in the uterine cavity exceeds 10 mm on ultrasonography and is accompanied by the presence of clinical symptoms such as vaginal bleeding and abdominal pain .The other type of miscarriage is defined as retained products of conception (RPOC) and refers to the state when the gestational sac contains the embryo with crown-rump length (CRL) of > 7 mm but embryonic cardiac activity is invisible. Empty gestational sac is diagnosed when the gestational sac with a diameter of > 25 mm and without an embryo is visible in the uterine cavity on ultrasonography .

Histopathological examination of products of conception is an integral and a routine component of the management of patients with early pregnancy failure . Two important primary reasons for such an examination are to confirm the presence of an intrauterine gestation and to exclude gestational trophoblastic disease in the form of partial or complete hydatidiform mole .

ELIGIBILITY:
Inclusion Criteria:

* all pregnants with clinical symptoms and signs of abortion
* fit for medical induction of abortion
* fit for surgical procedure

Exclusion Criteria:

* threatened abortion
* complete abortion
* unfit participants for medical abortion
* unfit participants for surgical procedure

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — All of the patients had vaginal bleeding and pelvic pain. After vaginal examination , transvaginal ultrasonography findings and serum β-HCG levels were performed to verify the diagnosis. The cases were classified as complete, incomplete, missed, or anembryonic miscarriage according to the guidelines of the Royal College of Obstetrics and Gynecology (RCOG) on the basis of transvaginal ultrasonography[5].
  Missed miscarriage was defined as the presence of a non-viable fetus. An intact gestational sac with an absence of fetal echo was diagnosed as an anembryonic miscarriage. Incomplete miscarriage was defined as the presence of heterogeneous tissues (with or without a gestational sac) distorting the endometrial midline echo by transvaginal ultrasonography.
Enrollment: 300 (Estimated)
Dates: Start 2020-12-20 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
percentage of results of products of conception assessed by histopathological evaluation | one year
  to asses the result of analysis of products of abortion and divide them into groups according to the results and asses percentage of each type types predicted :1-products of conception 2-no products of conception 3-partial moel 4-complete mole 5-Arias-stella reaction 6-others

SECONDARY OUTCOMES:
rate of participants show chronic histiocytic intervillositis in histopathological evaluation | one year
  assesment of chronic histiocytic intervillositis by detection of massive perivillous histiocytosis in placental tissue by histopathological evaluation

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Poland BJ, Miller JR, Jones DC, Trimble BK. Reproductive counseling in patients who have had a spontaneous abortion. Am J Obstet Gynecol. 1977 Apr 1;127(7):685-91. doi: 10.1016/0002-9378(77)90240-x. PMID 848521
- [Background] WARBURTON D, FRASER FC. SPONTANEOUS ABORTION RISKS IN MAN: DATA FROM REPRODUCTIVE HISTORIES COLLECTED IN A MEDICAL GENETICS UNIT. Am J Hum Genet. 1964 Mar;16(1):1-25. No abstract available. PMID 14131871
- [Background] Doubilet PM, Benson CB, Bourne T, Blaivas M; Society of Radiologists in Ultrasound Multispecialty Panel on Early First Trimester Diagnosis of Miscarriage and Exclusion of a Viable Intrauterine Pregnancy; Barnhart KT, Benacerraf BR, Brown DL, Filly RA, Fox JC, Goldstein SR, Kendall JL, Lyons EA, Porter MB, Pretorius DH, Timor-Tritsch IE. Diagnostic criteria for nonviable pregnancy early in the first trimester. N Engl J Med. 2013 Oct 10;369(15):1443-51. doi: 10.1056/NEJMra1302417. No abstract available. PMID 24106937
- [Background] Lemmers M, Verschoor MAC, Bossuyt PM, Huirne JAF, Spinder T, Nieboer TE, Bongers MY, Janssen IAH, Van Hooff MHA, Mol BWJ, Ankum WM, Bosmans JE; MisoREST study group. Cost-effectiveness of curettage vs. expectant management in women with an incomplete evacuation after misoprostol treatment for first-trimester miscarriage: a randomized controlled trial and cohort study. Acta Obstet Gynecol Scand. 2018 Mar;97(3):294-300. doi: 10.1111/aogs.13283. Epub 2018 Jan 19. PMID 29266169
- [Background] Luise C, Jermy K, May C, Costello G, Collins WP, Bourne TH. Outcome of expectant management of spontaneous first trimester miscarriage: observational study. BMJ. 2002 Apr 13;324(7342):873-5. doi: 10.1136/bmj.324.7342.873. PMID 11950733